CLINICAL TRIAL: NCT06791538
Title: A Multicenter, Prospective, Randomized Controlled Clinical Study of Robotic Versus Laparoscopic Radical Surgery for Locally Advanced Gastric Cancer
Brief Title: Robotic Versus Laparoscopic Radical Surgery for Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yan Shi, Chief Physician, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYRL-01
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer
Keywords: Robotic Gastrectomy; Laparoscopic Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Gastrectomy (Experimental)
  Interventions: Procedure: Robotic Gastrectomy
- Laparoscopic Gastrectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic Gastrectomy

INTERVENTIONS:
Procedure: Robotic Gastrectomy — The intervention measures for robotic gastrectomy include:
  Preoperative Preparation: Comprehensive preoperative examinations, including imaging studies, laboratory tests, and tumor marker assessments, to confirm the diagnosis and staging.
  Surgical Procedure: Utilizing the da Vinci Surgical System, which provides a high-definition 3D view and flexible robotic arms for enhanced surgical precision.
  Lymphadenectomy: Systematic D2 lymph node dissection according to oncological standards to ensure thorough removal of regional lymph nodes.
  Gastrectomy and Reconstruction: Performing subtotal or total gastrectomy based on tumor location and extent, with intracorporeal reconstruction assisted by the robotic system.
  Postoperative Management: Close monitoring of vital signs, pain management, and early mobilization to facilitate recovery, along with prevention and management of postoperative complications.
  Arms: Robotic Gastrectomy
Procedure: Laparoscopic Gastrectomy — Preoperative Preparation: Confirm diagnosis and staging through imaging and laboratory tests.
  Surgical Procedure: Use standard laparoscopic instruments and 2D HD camera. Lymphadenectomy: Perform systematic D2 lymph node dissection. Gastrectomy and Reconstruction: Conduct subtotal or total gastrectomy and intracorporeal reconstruction.
  Postoperative Management: Monitor vital signs, manage pain, and promote early mobilization.
  Arms: Laparoscopic Gastrectomy

SUMMARY:
This [Study Type: Clinical Trial] aims to [Primary Objective: evaluate the long-term efficacy and safety of robotic gastrectomy for locally advanced gastric cancer] in [Participant Population: patients with locally advanced gastric cancer, aged >18 years and <75 years]. The primary questions it seeks to answer are:

Is the 3-year disease-free survival rate of robotic gastrectomy non-inferior to that of laparoscopic gastrectomy? Is the perioperative safety of robotic gastrectomy superior to that of laparoscopic gastrectomy? Researchers will compare [Intervention Groups: Robotic Gastrectomy vs. Laparoscopic Gastrectomy] to determine whether [robotic surgery offers advantages in long-term efficacy and perioperative safety].

Participants will:

Sign an informed consent form and be randomly assigned to either the robotic surgery group or the laparoscopic surgery group.

Undergo the assigned surgical procedure and receive regular follow-up visits (at 30 days, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 2 years, 2.5 years, and 3 years postoperatively).

Complete physical examinations, blood tests (including complete blood count, biochemical markers, and tumor markers), and imaging studies (such as abdominal CT, upper gastrointestinal endoscopy, and chest X-ray) during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years and < 75 years.
2. Primary gastric lesion histologically confirmed as gastric adenocarcinoma (including papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, poorly differentiated adenocarcinoma, etc.) via endoscopic biopsy.
3. Preoperative clinical staging as locally advanced gastric cancer (cT2-4a, N0-3, M0) according to the 8th edition of the AJCC TNM staging system.
4. No distant metastasis on preoperative examination, and no direct invasion of the pancreas, spleen, or other adjacent organs.
5. Preoperative ECOG performance status score of 0 or 1.
6. Preoperative ASA (American Society of Anesthesiologists) physical status score of I-III.
7. Consent to participate in the study and signing of the informed consent form.

Exclusion Criteria:

1. Previous history of gastric malignancy surgery, including submucosal resection and/or endoscopic mucosal resection.
2. History of upper abdominal surgery (excluding laparoscopic cholecystectomy).
3. Preoperative imaging shows regional lymph nodes with confluent enlargement (maximum diameter ≥3cm).
4. Patient underwent emergency surgery due to gastric tumor bleeding or perforation.
5. History of other malignancies, or presence of other malignant tumors detected during preoperative examination.
6. Patient has a history of malignant tumor, or other malignant tumors were found during preoperative examination
7. ASA (American Society of Anesthesiologists) score >3.
8. Severe psychiatric disorders.
9. History of unstable angina or myocardial infarction within the past 6 months.
10. History of cerebral infarction or cerebral hemorrhage within the past 6 months.
11. Severe pulmonary disease with FEV1 < 50%.
12. Systemic corticosteroid therapy within 1 month prior to the study.
13. Need for concurrent surgery for other diseases.
14. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | 3 years

SECONDARY OUTCOMES:
Overall postoperative complication rate | 3 years
Intraoperative complication rate | 3 years
Overall postoperative complication rate of Clavien-Dindo Grade II or higher | 3 years
3-year OS rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Southwest hospital of AMU, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No